CLINICAL TRIAL: NCT00003753
Title: A Phase I-II Study of Hepatic Arterial Therapy Via Pump (Protocol D97-063) With Floxuridine (FUDR) and Dexamethasone (DEX) in Combination With Intravenous Irinotecan as Adjuvant Treatment After Resection of Hepatic Metastases From Colorectal Cancer
Brief Title: Floxuridine, Dexamethasone, and Irinotecan After Surgery in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 98-072; CDR0000066876 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-98072A(9); NCI-H99-0024
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Dexamethasone; Floxuridine; Irinotecan; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: dexamethasone
Drug: floxuridine
Drug: irinotecan hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as floxuridine, dexamethasone, and irinotecan, use different ways to stop tumor cells from dividing so they stop growing or die. Hepatic arterial infusion uses a catheter to deliver chemotherapy directly to the liver. Combining more than one drug and giving them in different ways may kill any tumor cells remaining after surgery.

PURPOSE: Phase II trial to study the effectiveness of irinotecan combined with hepatic arterial infusion with floxuridine and dexamethasone after surgery in treating patients who have liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of hepatic arterial infusion of floxuridine (FUDR) and dexamethasone given via an implanted pump in combination with weekly intravenous irinotecan as adjuvant treatment after resection of hepatic metastases in patients with hepatic metastases from colorectal cancer. (The MTDs of irinotecan and floxuridine have been reached as of 10/15/03; phase I closed to accrual as of 10/15/03.)
* Determine the efficacy of this combination chemotherapy after liver resection, in terms of 2-year survival and 2-year recurrence rates, in these patients.
* Determine the pharmacokinetic effects of intrahepatic FUDR and liver resection on the metabolism of irinotecan to its active metabolite, SN-38 in these patients.
* Determine the safety and efficacy of the pump used in delivering intra-arterial chemotherapy to the liver in these patients.

OUTLINE: This is a dose-escalation* study of floxuridine and irinotecan.

Patients undergo hepatic resection and pump placement into the abdomen. About 4 weeks after surgery, patients receive irinotecan IV over 30 minutes on days 1 and 15. Patients also receive floxuridine and dexamethasone intra-arterially via an implanted pump continuously on days 1-14. Treatment repeats every 28 days for 6 courses in the absence of unacceptable toxicity or disease progression.

Sequential dose escalation of irinotecan is followed by sequential dose escalation of floxuridine. Cohorts of 3-6 patients receive escalating doses of irinotecan and floxuridine until the maximum tolerated doses (MTDs) are determined. The MTD* (phase II dose) is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

NOTE: *The MTDs of irinotecan and floxuridine have been reached as of 10/15/03; phase I closed to accrual as of 10/15/03

Patients are followed every 3 months for 2 years, every 4 months for 2-4 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 2-24 patients will be accrued for the phase I portion of this study within 1 year (phase I closed to accrual as of 10/15/03). A total of 50 additional patients will be accrued for this study at the phase II dose level.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma
* Primary colorectal tumor must have been previously resected
* Potentially completely resectable hepatic metastases (or removable by cryoresection) without current evidence of other metastatic disease
* No extrahepatic sites of disease
* No ascites or hepatic encephalopathy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the liver
* At least 4 weeks since prior radiotherapy to the pelvis

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Kemeny, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States